CLINICAL TRIAL: NCT01738724
Title: Abnormal Uterine Bleeding in Women With Uterine Leiomyomas: Open Randomized Clinical Trial Of Non Inferiority Between Oral Dienogest, Oral Desogestrel and Subcutaneous Goserelin
Brief Title: Study of the Efficacy of Dienogest in the Treatment of Uterine Leiomyomas When Compared to Desogestrel and Goserelin
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI went for a post-doc course and when he came back he moved for another job
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, LUIZ GUSTAVO OLIVEIRA BRITO, Assistant Physician, MD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMRPUSP-UROGIN-002
Record Dates: First submitted 2012-11-23; First posted 2012-11-30 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Uterine Leiomyoma
MeSH Terms: conditions — Myofibroma | interventions — dienogest; Goserelin; Desogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dienogest (Experimental): Dienogest 2mg pills daily during 6 months
  Interventions: Drug: Dienogest
- Goserelin (Experimental): Goserelin 10.8mg preloaded syringe subcutaneously at the start of the study and after 3 months
  Interventions: Drug: Goserelin
- Desogestrel (Active Comparator): Desogestrel 75mcg pills daily during six months
  Interventions: Drug: Desogestrel

INTERVENTIONS:
Drug: Dienogest — Dienogest 2mg pills daily during 6 months
  Other Names: Allurene; Visanne
  Arms: Dienogest
Drug: Goserelin — Goserelin 10.8mg preloaded syringe subcutaneously at the start of the study and after 3 months
  Other Names: Zoladex
  Arms: Goserelin
Drug: Desogestrel — Desogestrel 75mcg pills daily during six months
  Other Names: Cerazette
  Arms: Desogestrel

SUMMARY:
The investigators´aim is to assess whether the progestagen dienogest reduces leiomyoma volume and its associated symptoms to the same extent as gonadotropin releasing hormone (GnRH) analogs or the progestagen desogestrel or whether it is inferior to other drugs already in use.

DETAILED DESCRIPTION:
Uterine leiomyoma is a very prevalent condition among women and, although it is mainly asymptomatic, it may be related to bothersome or debilitating symptoms, such as uterine bleeding and pelvic pain or pressure. The standard treatment is surgical (hysterectomy or myomectomy), but there has been continued interest on medical treatments. Progestagens have long been used to control bleeding associated to leiomyomas, but they have not been able to decrease myoma volume. GnRH analogs are well stablished agents, capable of controlling symptoms and decreasing the tumors´volume, but their use is limited by bone loss and menopausal symptoms. A newly introduced progestagen, dienogest, has been studied to treat endometriosis, but its effects on leiomyoma are only starting to be assessed. The investigators are aiming to compare dienogest with the GnRH analog goserelin and the progestagen desogestrel in a randomized trial to see how this new treatment compares with previously used drugs and whether it is similar, inferior or superior to them on controlling leiomyoma associated symptoms and decreasing leiomyoma volume.

ELIGIBILITY:
Inclusion Criteria:

* Women with 35 - 55 years of age
* Uterine volume between 50cc and 500cc
* Abnormal uterine bleeding probably associated to intramural uterine leiomyomas

Exclusion Criteria:

* Pregnancy
* Liver or kidney dysfunction
* Women with only submucosal or subserosal uterine leiomyomas
* Women with contraindications to any of the drugs (categories 3 and 4 of WHO eligibility criteria)
* Use of anticoagulants
* Others causes of abnormal uterine bleeding (endometrial pathology, cervical pathology)

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Leiomyoma Volume | After 6 months of medical therapy

SECONDARY OUTCOMES:
Pictorial Blood Assessment Chart (PBAC) Score Reduction | After 6 months of medical therapy
Number of episodes of vaginal bleeding | After 6 months of medical therapy

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Gustavo O Brito, MD, PhD, Study Chair — FMRP-USP